CLINICAL TRIAL: NCT01179620
Title: A Multi-center, Prospective, Open-label, 8-weeks Study to Investigate the Efficacy, Safety and Pharmacokinetics of Certoparin (3000 IU Anti-Xa Bolus, With the Option to Titrate Dose)in the Prophylaxis of Clotting in the Extracorporeal Circuit in Patients Undergoing Chronic Hemodialysis
Brief Title: Certoparin in Renal Patients Undergoing Hemodialysis
Acronym: MEMBRANE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CMEX839BDE06
Record Dates: First submitted 2010-07-27; First posted 2010-08-11 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Renal Dialysis
Keywords: Hemodialysis, Certoparin
MeSH Terms: interventions — certoparin

ARMS (1):
- Certoparin (Experimental)
  Interventions: Drug: Certoparin

INTERVENTIONS:
Drug: Certoparin — Certoparin

SUMMARY:
This study will assess the efficacy, safety and pharmacokinetics of certoparin when used to prevent clotting during hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring hemodialysis
* Patients requiring anticoagulation therapy during hemodialysis
* Written informed consent

Exclusion Criteria:

* Hypersensitivity to study medication
* Genetic abnormality or disease of clotting system
* Prior major surgery or bleeding
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Number of patients requiring uptitration | Week 8

SECONDARY OUTCOMES:
Pharmacokinetics of Certoparin | Day 1, Week 4
Safety and tolerability of Certoparin | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Germany (9):
  - Novartis Investigative Site Darmstadt, Darmstadt
  - Novartis Investigative Site Elsenfeld, Elsenfeld
  - Novartis Investigative Site Flensburg, Flensburg
  - Novartis Investigative Site Heringen, Heringen
  - Novartis Investigative Site Hoyerswerda,, Hoyerswerda
  - Novartis Investigative Site Kronach, Kronach
  - Novartis Investigative Site Magdeburg, Magdeburg
  - Novartis Investigative Site München, München
  - Novartis Investigative Site Münster, Münster

REFERENCES:
- [Derived] Dorsch O, Krieter DH, Lemke HD, Fischer S, Melzer N, Sieder C, Bramlage P, Harenberg J. A multi-center, prospective, open-label, 8-week study of certoparin for anticoagulation during maintenance hemodialysis--the membrane study. BMC Nephrol. 2012 Jun 28;13:50. doi: 10.1186/1471-2369-13-50. PMID 22742742